

#### Protocol C2321005

A Phase 1, Randomized, Open-label, 3-period, crossover, single-dose, 2-part study in healthy participants to investigate the effect of tablet formulation and food on the relative bioavailability of PF-06821497

Statistical Analysis Plan (SAP)

Version: 1

**Date:** 30 Mar 2023

# TABLE OF CONTENTS

| LIST OF TABLES | 4 |
|-------------------------------------------------------------------|----|
| APPENDICES | 4 |
| 1. VERSION HISTORY | 5 |
| 2. INTRODUCTION | 5 |
| 2.1. Modifications to the Analysis Plan Described in the Protocol | 5 |
| 2.2. Study Objectives and Endpoints | 5 |
| 2.3. Study Design | 6 |
| 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 8 |
| 3.1. Primary Endpoints | 8 |
| 3.2. Secondary Endpoints | 8 |
| 3.3. Baseline Variables | 8 |
| 3.4. Other Endpoints | 8 |
| 3.5. Safety Endpoints | 9 |
| 3.5.1. Adverse Events | 9 |
| 3.5.2. Laboratory Data | 10 |
| 3.5.3. Vital Signs | 10 |
| 3.5.4. Electrocardiograms. | 10 |
| 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS) | 10 |
| 5. GENERAL METHODOLOGY AND CONVENTIONS | 11 |
| 5.1. Hypotheses and Decision Rules | 11 |
| 5.2. General Methods | 11 |
| 5.2.1. Analyses for Binary/Categorical Endpoints | 11 |
| 5.2.2. Analyses for Continuous Endpoints | 11 |
| 5.3. Methods to Manage Missing Data | 11 |
| 5.3.1. Pharmacokinetic Data | 11 |
| 5.3.2. Safety Data | 12 |
| 6. ANALYSES AND SUMMARIES | 13 |
| 6.1. Primary Endpoints | 13 |
| 6.2. Secondary Endpoints | 13 |
| 6.3. Other Endpoints | 14 |

| 6.4. Subset Analyses | 15 |
|-------------------------------------------------------|----|
| 6.5. Baseline and Other Summaries and Analyses | 15 |
| 6.5.1. Demographic Summaries | 15 |
| 6.5.2. Study Conduct and Participant Disposition | 16 |
| 6.5.3. Study Treatment Exposure | 16 |
| 6.5.4. Concomitant Medications and Nondrug Treatments | 16 |
| 6.6. Safety Summaries and Analyses | 16 |
| 6.6.1. Adverse Events | 16 |
| 6.6.2. Laboratory Data | 16 |
| 6.6.3. Vital Signs | 16 |
| 6.6.4. Electrocardiograms | 16 |
| 7. INTERIM ANALYSES | 16 |
| APPENDICES | 17 |

## LIST OF TABLES

| Table 1. | Summary of Changes | 5 |
|---|---|---|
| Table 2. | Treatment Schedule | 7 |
| Table 3. | Plasma PF-06821497 PK Parameters Definitions | 9 |
| Table 4. | PK Parameters to be Summarized Descriptively by Treatment | 14 |
| | APPENDICES | |
| Appendix 1. S | SAS Code for Analyses | 17 |
| Appendix 2. 1 | List of Abbreviations | 19 |

NOTE: Italicized text within this document has been taken verbatim from the Protocol.

#### 1. VERSION HISTORY

**Table 1. Summary of Changes** 

| Version/<br>Date | Associated Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1 /<br>30 Mar 2023 | Original<br>02 Feb 2023 | N/A | N/A |

#### 2. INTRODUCTION

PF-06821497 is a potent and selective inhibitor of EZH2 as evidenced by its biochemical inhibition of both WT and EZH2 Y641N mutant enzymes. PF-06821497 is currently being proposed for investigation in patients with SCLC, CRPC, DLBCL, and FL.

The purpose of the study is to investigate the relative bioavailability of tablet formulations of PF-06821497 and to characterize the effect of food on a PF-06821497 tablet formulation (Formulation 2). The data generated from this study will be used to support the pivotal study formulation, to inform dose administration instructions for PF-06821497 with regard to dosing with or without food, and to enable the establishment of the API particle size specifications for eventual commercialization.

This SAP provides the detailed methodology for summary and statistical analyses of the data collected in Study C2321005.

## 2.1. Modifications to the Analysis Plan Described in the Protocol

None.

## 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary: | Primary: |
| To estimate the bioavailability of a single of mg dose of PF-06821497 tablet formulation (Formulation 2) relative to a single mg dose of PF-06821497 tablet formulation (Formulation 1) under fasted conditions in adult healthy participants | • Plasma AUC <sub>inf</sub> and C <sub>max</sub> for PF-06821497. (AUC <sub>last</sub> will be used as the primary estimate if AUC <sub>inf</sub> cannot be reliably estimated). |
| Secondary: | Secondary: |
| • To estimate the bioavailability of a single mg dose of PF-06821497 tablet (larger API particle size) formulation (Formulation 3) relative to a single mg dose of PF-06821497 tablet (Formulation 2) and a single 250 mg dose of the PF-06821497 tablet formulation (Formulation 1) under fasted conditions in adult healthy participants | • Plasma AUC <sub>inf</sub> and C <sub>max</sub> for PF-06821497 for tablet (larger API particle size) (Formulation 3) relative to (Formulation 2) and tablet (Formulation 1) formulations. (AUC <sub>last</sub> will be used as the primary estimate if AUC <sub>inf</sub> cannot be reliably estimated). |

| Objectives | Endpoints |
|---|---|
| • To estimate the effect of a high-fat, high-calorie meal on the bioavailability of a single of mg dose of the PF-06821497 tablet formulation (Formulation 2) relative to fasted conditions in adult healthy participants | • Plasma AUC <sub>inf</sub> and C <sub>max</sub> for PF-06821497 under fed (high-fat, high-calorie meal) conditions relative to fasting conditions. (AUC <sub>last</sub> will be used as the primary estimate if AUC <sub>inf</sub> cannot be reliably estimated). |
| To estimate the effect of a low-fat, low-calorie meal on the bioavailability of a single mg dose of the PF-06821497 tablet formulation (Formulation 2) relative to fasted conditions in adult healthy participants | • Plasma AUC <sub>inf</sub> and C <sub>max</sub> for PF-06821497 under fed (low-fat, low-calorie meal) conditions relative to fasting conditions. (AUC <sub>last</sub> will be used as the primary estimate if AUC <sub>inf</sub> cannot be reliably estimated). |
| To evaluate the safety and tolerability of PF-<br>06821497 when administered as a tablet<br>formulation to healthy participants | Assessment of TEAEs, clinical laboratory<br>abnormalities, vital signs, physical examinations,<br>and 12-lead ECGs. |

## 2.3. Study Design

This is a Phase 1, randomized, open-label, 3-period, crossover, single-dose 2-part study in healthy participants to investigate the effect of tablet formulation and food on the bioavailability of PF-06821497.

In each part of the study, each enrolled participant will participate in 3 study periods to receive 3 different treatments according to the sequence determined by randomization with 5-day washouts between PF-06821497 administration:

## *Part 1 (rBA)*:

- Treatment A Single of mg dose (Formulation (Formulation 1), under fasting conditions (following an overnight fast of at least 10 hours)
- Treatment B Single of mg dose of WG tablet formulation (Formulation 2), under fasting conditions (following an overnight fast of at least 10 hours)
- Treatment C Single of mg dose API particle size) (Formulation 3), under fasting conditions (following an overnight fast of at least 10 hours)

## Part 2 (Food Effect):

- Treatment D Single CCI tablet formulation (Formulation 2), under fasting conditions (following an overnight fast of at least 10 hours)
- Treatment E Single CCI tablet formulation (Formulation 2), given with a low-fat/low-calorie meal
- Treatment F Single  $\frac{|C|}{|C|}$  tablet formulation (Formulation 2), given with a high-fat/high-calorie meal

Approximately 18 participants will be enrolled to the study intervention. If there are participants who withdraw or discontinue treatment and are considered to be non-evaluable with respect to the primary PK objective(s), additional participants can be enrolled at the discretion of the investigator upon consulation with the sponsor.

In each part of the study, each enrolled participant will receive 1 of the 3 treatments in each period according to treatment schedule shown in Table 2.

**Table 2.** Treatment Schedule



# 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

## 3.1. Primary Endpoints

The primary endpoints are the plasma AUC<sub>inf</sub> (if data permit, otherwise AUC<sub>last</sub>) and C<sub>max</sub> for PF-06821497. The test/reference ratios for AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub> and C<sub>max</sub> will be derived with Treatment B ( formulation (Formulation 2) fasted) as the Test treatment and Treatment A ( formulation (Formulation 1) formulation (Formulation 1)

## 3.2. Secondary Endpoints

The test/reference ratios for AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub> and C<sub>max</sub> will be derived with Treatment C ( formulation (Formulation 3) ( larger API particle size) fasted) as the Test treatment and Treatment B ( formulation (Formulation 2) ( formulation 2) ( formulation 3) fasted) and Treatment A ( formulation (Formulation 1) ( formulation 1) ( formulation 3) ( formulation 4) ( formulation 3) ( formulation 4) ( formulation 3) ( formulation 4) ( formulation

The test/reference ratios for AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub> and C<sub>max</sub> will be derived with Treatments E and F ( formulation (Formulation 2) fed: low-fat meal and formulation (Formulation 2) fed: high-fat meal) as the Test treatments and Treatment D ( formulation (Formulation 2) formulation (Formulation 2) fested) as the Reference treatment.

Included as secondary endpoints are the safety and tolerability data, discussed in Section 3.5.

#### 3.3. Baseline Variables

Baseline characteristics will be collected according to the schedule of activities (SoA) as specified in the protocol.

#### 3.4. Other Endpoints

CCI

Plasma PK parameters of PF-06821497 will be derived (as data permits) from the concentration-time data using standard noncompartmental methods as outlined in Table 3. The PF-06821497 plasma PK parameters will be summarized descriptively by Treatment. Plasma concentrations will be listed and summarized descriptively by Treatment, and nominal PK sampling time. Individual participant and summary profiles (mean and median plots) of the plasma concentration time data will be plotted using actual and nominal times, respectively.

Actual PK sampling times will be used in the derivation of PK parameters. In the case that actual PK sampling times are not available, nominal PK sampling time will be used in the derivation of PK parameters.

Parameter Definition Method of Determination AUC<sub>inf</sub>\*  $AUC_{last} + (C_{last}*/k_{el}),$ area under the concentration-time curve from time 0 to infinity where  $C_{last}$ \* is the predicted plasma concentration at the last quantifiable time point from the loglinear regression analysis and  $k_{el}$  is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve  $AUC_{last}$ area under the concentration-time curve from 0 to Linear/Log trapezoidal method. time of last measurable concentration Observed directly from data  $C_{max}$ maximum observed concentration CC

Table 3. Plasma PF-06821497 PK Parameters Definitions

## 3.5. Safety Endpoints

The following data are considered in standard safety summaries (see protocol for collection days, baseline assessment, and list of parameters):

- adverse events (AE)
- laboratory data
- vital signs data
- electrocardiogram (ECG) results

#### 3.5.1. Adverse Events

Any adverse events occurring following start of treatment will be considered as treatment emergent adverse event (TEAE). Events that occur during follow-up within the lag time of up to 35 days after the last dose of study intervention will be counted as treatment emergent and attributed to the last treatment taken. The time period for collecting AEs ("active collection period") for each participant begins from the time the participant provides informed consent.

<sup>\*</sup>If data permits.

## 3.5.2. Laboratory Data

Safety laboratory tests will be performed as described in the protocol. To determine if there are any clinically significant laboratory abnormalities, the haematological, clinical chemistry (serum) and urinalysis safety tests will be assessed against the criteria specified in the sponsor reporting standards. The assessment will not take into account whether each participants's baseline test result is within or outside the laboratory reference range for the particular laboratory parameter.

For each period, the baseline measurement is the predose measurement on Day -1.

## 3.5.3. Vital Signs

Supine blood pressure (BP), pulse rate (PR), respiratory rate and temperature will be measured at times specified in the SoA given in the protocol.

For each period, the baseline measurement is the predose measurement on Day 1.

## 3.5.4. Electrocardiograms

QT interval, QTcF, PR interval, QRS and heart rate (HR) will be recorded at each assessment time indicated in the SoA given in the protocol. QTcF will be derived using Fridericia's heart rate correction formula:

QTcF = QT / 
$$(RR)^{(1/3)}$$
 where RR = 60/HR (if not provided)

For each period, the baseline measurement is the predose measurement on Day 1.

## 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS)

Data for all participants will be assessed to determine if participants meet the criteria for inclusion in each analysis population prior to releasing the database and classifications will be documented per standard operating procedures.

| Participant Analysis Set | Description |
|---|---|
| Enrolled | "Enrolled" means a participant's, or their legally authorized representative's, agreement to participate in a clinical study following completion of the informed consent process and assignment to study intervention. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. |

| Participant Analysis Set | Description |
|---|---|
| PK Concentration Population | The PK concentration population is defined as all participants randomized and treated who have at least 1 PF-06821497 concentration in at least 1 treatment period. |
| PK Parameter Population | The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the PF-06821497 PK parameters of primary interest in at least 1 treatment period. |
| Safety analysis set | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants will be analyzed according to the product they actually received. |

#### 5. GENERAL METHODOLOGY AND CONVENTIONS

Final analysis will be performed after study participant data set release following last participant last visit.

## 5.1. Hypotheses and Decision Rules

No statistical hypothesis will be tested in this study.

#### 5.2. General Methods

## 5.2.1. Analyses for Binary/Categorical Endpoints

For binary or categorical variables, number of participants, numbers and percentages of participants meeting the categorical criteria will be presented in accordance with the Clinical Data Interchange Standards Consortium and Pfizer Standards (CaPS).

#### **5.2.2.** Analyses for Continuous Endpoints

For continuous variables, the data will be summarized using the number of participants, mean, median, standard deviation (SD), minimum, and maximum in accordance with the CaPS. For appropriate PK parameters, geometric mean and geometric coefficient of variation (%CV) will also be summarized.

#### 5.3. Methods to Manage Missing Data

#### 5.3.1. Pharmacokinetic Data

Methods to handle missing PK data are described below.

## **Concentrations Below the Limit of Quantification:**

In all data presentations (except listings), concentrations below the limit of quantification (BLQ) will be set to zero. In listings, BLQ values will be reported as "<LLQ", where LLQ will be replaced with the value for the lower limit of quantification.

## **Deviations, Missing Concentrations and Anomalous Values:**

In summary tables and plots of median profiles, statistics will be calculated having set concentrations to missing if 1 of the following cases is true:

- 1. A concentration has been collected as ND (ie, not done) or NS (ie, no sample).
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged anomalous by the pharmacokineticist.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing.

An anomalous concentration value is one that, after verification of bioanalytical validity, is grossly inconsistent with other concentration data from the same individual or from other participants. For example, a BLQ concentration that is between quantifiable values from the same dose is considered as anomalous. Anomalous concentration values may be excluded from PK analysis at the discretion of the PK analyst.

#### **PK Parameters:**

Actual PK sampling times will be used in the derivation of PK parameters. If a PK parameter cannot be derived from a participant's concentration data, the parameter will be coded as NC (ie, not calculated). (Note that NC values will not be generated beyond the day that a participant discontinues).

In summary tables, statistics will not be presented for a particular treatment group if more than 50% of the data are NC. For statistical analyses, PK parameters coded as NC will also be set to missing.

If an individual participant has a known biased estimate of a PK parameter (due for example to a dosing error or an unexpected event such as vomiting before all the compound is adequately absorbed from the gastrointestinal tract), this will be footnoted in summary tables and will not be included in the calculation of summary statistics or statistical analyses.



## 5.3.2. Safety Data

Missing values in standard summaries of AEs and laboratory data will be imputed according to CaPS.

#### 6. ANALYSES AND SUMMARIES

### 6.1. Primary Endpoints

AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub> and C<sub>max</sub> will be summarized by treatment group and will include the set of summary statistics as specified in Table 4.

For the evaluation of relative bioavailability, natural log transformed  $AUC_{inf}$  (if data permit),  $AUC_{last}$  and  $C_{max}$  will be analyzed using a mixed effects model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals will be obtained from the model. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. Treatment A (CCI) formulation (Formulation 1) (CCI) fasted) will be the Reference treatment and Treatment B (CCI) formulation (Formulation 2) (CCI) fasted) will be the Test treatment.

For  $AUC_{inf}$ ,  $AUC_{last}$  and  $C_{max}$ , a listing of the individual participant ratios (Test/Reference) will be provided. Box and whisker plots for  $AUC_{inf}$ ,  $AUC_{last}$  and  $C_{max}$ , will be plotted by treatment and overlaid with geometric means.

Residuals from the model will be examined for normality and the presence of outliers via visual inspection of plots of residuals vs predicted values and normal probability plots of residuals but these will not be included in the CSR. If there are major deviations from normality or outliers then the effect of these on the conclusions will be investigated through alternative transformations and/or analyses excluding outliers. Justification for any alternative to the planned analysis will be given in the report of the study.

#### 6.2. Secondary Endpoints

For the evaluation of relative bioavailability, natural log transformed AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub> and C<sub>max</sub> will be analyzed using a mixed effects model with sequence and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals will be obtained from the model. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. Treatment A (CCI) formulation (Formulation 1) and pasted) will be the Reference treatment and Treatment C (CCI) formulation (Formulation 3) and pasted) will be the Reference treatment B (CCI) formulation (Formulation 2) and pasted) will be the Reference treatment and Treatment C (CCI) formulation (Formulation 3) and pasted treatment and Treatment C (CCI) formulation (Formulation 3) and pasted treatment and Treatment C (CCI) formulation (Formulation 3) and pasted treatment and Treatment C (CCI) formulation (Formulation 3) and pasted treatment and Treatment C (CCI) formulation (Formulation 3) and pasted treatment C (CCI) formulation (Formulation 3) and pasted treatment C (CCI) formulation (Formulation 4) and pasted treatment C (CCI) formulation (Formulation 4) and pasted treatment C (CCI) formulation (Formulation 4) and pasted treatment C (CCI) form

For the evaluation of food effect, natural log transformed  $AUC_{inf}$  (if data permit),  $AUC_{last}$  and  $C_{max}$  will be analyzed using a mixed effects model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference)

and corresponding 90% confidence intervals will be obtained from the model. The adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. Treatment D ( formulation (Formulation 2) formulation (Formulation 2) formulation (Formulation 2) formulation (Formulation 2) fed: high-fat meal) will be the Test treatments.

For AUC<sub>inf</sub>, AUC<sub>last</sub> and C<sub>max</sub>, a listing of the individual participant ratios (Test/Reference) will be provided. Box and whisker plots for AUC<sub>inf</sub>, AUC<sub>last</sub> and C<sub>max</sub>, will be plotted by treatment and overlaid with geometric means.

Residuals from the model will be examined for normality and the presence of outliers via visual inspection of plots of residuals vs predicted values and normal probability plots of residuals but these will not be included in the CSR. If there are major deviations from normality or outliers then the effect of these on the conclusions will be investigated through alternative transformations and/or analyses excluding outliers. Justification for any alternative to the planned analysis will be given in the report of the study.

Analyses and summaries of safety data are described in Section 6.6.

## 6.3. Other Endpoints

#### **PK Parameters:**

The PK parameters will be listed and summarized descriptively by treatment group in accordance with Pfizer data standards on the PK Parameter Analysis Set, as data permit. Missing values will be handled as detailed in Section 5.3.1. Each PK parameter will be summarized by treatment group and will include the set of summary statistics as specified in Table 4.

Table 4. PK Parameters to be Summarized Descriptively by Treatment

| Parameter | Summary Statistics |
|---|---|
| AUC <sub>inf</sub> , AUC <sub>last</sub> , C <sub>max</sub> , | N, arithmetic mean, median, SD, %CV, minimum, maximum, |
| CCI | geometric mean and geometric %CV |
| CCI | |

Supporting data from the estimation of  $t_{1/2}$  and  $AUC_{inf}$  will be listed by analyte and group: terminal phase rate constant ( $k_{el}$ ); goodness of fit statistic from the log-linear regression ( $r^2$ ); the percent of  $AUC_{inf}$  based on extrapolation ( $AUC_{extrap}$ %); and the first, last, and number of time points used in the estimation of  $k_{el}$ . This data may be included in the clinical study report.

#### **PK Concentrations:**

The plasma concentrations will be listed and descriptively summarized by nominal PK sampling time and treatment. Individual participant, as well as mean and median profiles of the plasma concentration time data will be plotted by treatment using actual (for individual) and nominal (for mean and median) times respectively. Mean and median profiles will be presented on both linear and semi-log scales.

Presentations of concentrations will include:

- A listing of all concentrations sorted by participant ID, treatment and nominal time postdose. The concentration listing will also include the actual times. Deviations from the nominal time will be given in a separate listing.
- A summary of concentrations by treatment and nominal time postdose, where the set of statistics will include n, mean, median, SD, %CV, minimum, maximum and the number of concentrations above the LLQ.
- Median concentrations time plots (on both linear and semi-log scales) against nominal time postdose by treatment (all treatments on the same plot per scale, based on the summary of concentrations by treatment and time postdose).
- Mean concentrations time plots (on both linear and semi-log scales) against nominal time postdose by treatment (all treatments on the same plot per scale, based on the summary of concentrations by treatment and time postdose).
- Individual concentration time plots by treatment (on both linear and semi-log scales) against actual time postdose (there will be separate spaghetti plots for each treatment per scale).

Individual concentration time plots by participant (on both linear and semi-log scales) against actual time postdose [there will be separate plots for each participant (containing all treatments) per scale].

#### **6.4. Subset Analyses**

There are no planned subset analyses.

#### 6.5. Baseline and Other Summaries and Analyses

#### 6.5.1. Demographic Summaries

Demographic characteristics will be summarized for enrolled population in accordance with the CaPS.

## 6.5.2. Study Conduct and Participant Disposition

Participants evaluation groups will show end of study participant disposition. Frequency counts will be supplied for participant discontinuation(s) by treatment. Data will be reported in accordance with the CaPS.

## 6.5.3. Study Treatment Exposure

Study treatment exposure will be listed.

## 6.5.4. Concomitant Medications and Nondrug Treatments

All prior and concomitant medication(s) as well as non-drug treatment(s) will be reported in the listings.

## 6.6. Safety Summaries and Analyses

All safety analyses will be performed on the Safety Analysis Set.

Safety data will be presented in tabular and/or graphical format and summarized descriptively, where appropriate.

#### 6.6.1. Adverse Events

Adverse events will be reported in accordance with the CaPS.

Participant discontinuations due to adverse events will be detailed by treatment. Data will be reported in accordance with the CaPS.

#### 6.6.2. Laboratory Data

Laboratory data will be listed and summarized by treatment in accordance with the CaPS.

## 6.6.3. Vital Signs

Vital sign data will be databased and available upon request.

## 6.6.4. Electrocardiograms

ECG data will be databased and available upon request.

#### 7. INTERIM ANALYSES

No formal interim analysis will be conducted for this study. As this is an open-label study, the sponsor may conduct unblinded reviews of the data during the course of the study for the purpose of safety assessment, facilitating PK/PD modeling, and/or supporting clinical development.

Final analysis will follow the official database release. As this will be an open-label study, there is no formal unblinding of the randomization code.

#### **APPENDICES**

## **Appendix 1. SAS Code for Analyses**

An example of the PROC MIXED code is provided below:

## For the primary objective – relative BA:

```
proc mixed data=tab.pk;
    class seq period trt participant;
    model l&var=seq period trt/ ddfm=KR;
    random participant(seq) /subject=participant(seq);
    lsmeans trt;
    estimate 'B vs A' trt -1 1 0 /cl alpha=0.1;

    ods 'Estimates' out=est&var;
    ods 'Ismeans' out=ls&var;
    ods 'covparms' out=cov&var;
    ods 'tests3' out=tst&var;
run;
```

## For the secondary objective – relative BA:

```
proc mixed data=tab.pk;
       class seq trt participant;
       model 1&var=seq trt/ ddfm=KR;
       random participant(seq)/subject=participant(seq);
       1smeans trt;
       estimate 'C vs A' trt -1 0 1 /cl alpha=0.1;
       ods 'Estimates' out=est&var;
       ods 'lsmeans' out=ls&var;
       ods 'covparms' out=cov&var;
       ods 'tests3' out=tst&var;
run:
proc mixed data=tab.pk;
       class seq trt participant;
       model l&var=seq trt/ ddfm=KR;
       random participant(seq)/subject=participant(seq);
       lsmeans trt;
       estimate 'C vs B' trt 0 -1 1 /cl alpha=0.1;
       ods 'Estimates' out=est&var;
       ods 'lsmeans' out=ls&var;
       ods 'covparms' out=cov&var;
       ods 'tests3' out=tst&var;
run;
```

## For the secondary objective – food effect:

```
proc mixed data=tab.pk;
       class trt participant;
       model 1&var= trt/ ddfm=KR;
       random participant/subject=participant;
       1smeans trt;
       estimate 'E vs D' trt -1 1 0 /cl alpha=0.1;
       ods 'Estimates' out=est&var:
       ods 'lsmeans' out=ls&var;
       ods 'covparms' out=cov&var;
       ods 'tests3' out=tst&var;
run;
proc mixed data=tab.pk;
       class trt participant;
       model l&var= trt/ ddfm=KR;
       random participant/subject=participant;
       Ismeans trt;
       estimate 'F vs D' trt -1 0 1 /cl alpha=0.1;
       ods 'Estimates' out=est&var;
       ods 'lsmeans' out=ls&var;
       ods 'covparms' out=cov&var;
       ods 'tests3' out=tst&var;
run;
/* Letter assignments for treatments (trt) within the estimate statement above are as follows
Treatment A – CCI
                   formulation (Formulation 1)
                                                                      fasted;
               formulation (Formulation 3)
                  formulation (Formulation 2)
                                                                     fasted;
Treatment B –
                                                                     larger API particle
Treatment C –
size) fasted;
Treatment D – WG formulation (Formulation 2)
                                                                      fasted;
Treatment E – WG formulation (Formulation 2)
                                                                      fed: Low-fat meal;
Treatment F – WG formulation (Formulation 2)
                                                                      fed: High-fat meal */
```

# Appendix 2. List of Abbreviations

| Abbreviation | Term |
|---|---|
| %CV | coefficient of variation |
| AE | adverse event |
| API | Active Pharmaceutical Ingredients |
| AUC <sub>extrap</sub> % | the percent of AUC <sub>inf</sub> based on extrapolation |
| AUCinf | area under the concentration-time curve from time 0 to infinity |
| AUC <sub>last</sub> | area under the concentration-time curve from 0 to time of last measurable concentration |
| BA | bioavailability |
| BLQ | below the limit of quantitation |
| BP | blood pressure |
| CaPS | Clinical Data Interchange Standards Consortium and Pfizer Standards |
| CI | confidence interval |
| C <sub>last</sub> | last quantifiable concentration |
| CCI | • |
| C <sub>max</sub> | maximum observed concentration |
| CRPC | castration resistant prostate cancer |
| CSR | clinical study report |
| DLBCL | diffuse large B-cell lymphoma |
| ECG | electrocardiogram |
| FL | follicular lymphoma |
| HR | heart rate |
| kel | terminal phase rate constant |
| LLQ | lower limit of quantitation |
| mg | milligram |
| CCI | |
| N/A | not applicable |
| NC | not calculated |
| ND | not done |
| NS | no sample |
| PD | pharmacodynamic(s) |
| PK | pharmacokinetic(s) |
| PR | pulse rate |
| PR interval | time from the beginning of the P wave to the beginning of the QRS |
| | complex |
| QRS | Combination of Q-, R- and S- wave on an electrocardiogram representing |
| | ventricular depolarization |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |
| $r^2$ | goodness of fit statistic from the log-linear regression |
| rBA | relative bioequivalence |

| Abbreviation | Term |
|---|---|
| RR | the time between the start of one QRS complex and the start of the next |
| | QRS complex |
| SAP | statistical analysis plan |
| SCLC | small cell lung cancer |
| SD | single dose; standard deviation |
| SoA | schedule of activities |
| TEAE | treatment emergent adverse event |
| CCI | |
| WT | wild type |